CLINICAL TRIAL: NCT06775106
Title: Exhaled Breath: A Novel Technique for Rapid Diagnosis of Respiratory Diseases and Infections
Acronym: EXB
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Albert Chi, M.D., F.A.C.S., Oregon Health and Science University
Other Study IDs: 27461
Record Dates: First submitted 2024-08-27; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Disease; Critical Illness
Keywords: ventillator; critical care; pulmonary disease; inflammatory biomarkers
MeSH Terms: conditions — Lung Diseases; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-COVID patients on ventilator support: There is only one arm in the study, no randomization. Any non-COVID patient admitted to the ICU and requiring ventilation support will be eligible for enrollment into the study.
  Interventions: Other: There is no intervention in this observational study

INTERVENTIONS:
Other: There is no intervention in this observational study — No direct intervention will be done to patients eligible for the study. There will be a shunt placed to divert 5-15% of exhaled breath into a collection tube. This will not affect the patient's existing standard medical care.

SUMMARY:
This study aims to use mass spectrometry techniques to analyze exhaled patient breath in non-COVID ICU-admitted patients requiring ventilation for a rapid and accurate early detection of pulmonary diseases and inflammatory markers.

DETAILED DESCRIPTION:
The major aim of this observational study is to validate the new technique, Orbitrap and Matrix-Assisted Laser Desorption Ionization (MALDI) mass spectrometry, to sample and analyze exhaled patient breath that may be then used in non-intensive care unit (ICU) environments where rapid virus or other respiratory pathogen detection is of great utility. The ICU permits the direct measure of ventilator-dependent patients with known pulmonary disease (by sputum, chest x-ray, and/or bronchial lavage analysis) together with a simple, pure, and concentrated breath sample (expired air via ventilator tubing) for analysis.

Sub-aim 1: Run patient samples on Orbitrap & MALDI. Proteins in the samples will be captured and analyzed by Orbitrap and MALDI mass spectrometry. Selected proteins will be enzymatically digested into peptides and correlations to existing peptides from previous proteomic studies of exhaled breath condensates (EBC) will be examined. Candidate virus & bacterial proteins, as well as other cellular and biomarkers, will be cataloged.

Sub-aim 2: Correlate collected analyzed sample collection during hospitalization with other hospital data that may have been collected for clinical reasons by the clinical care team, at or around the study time period (+/- 3 days), concerning for the laboratory diagnosis of respiratory disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-COVID-19 adult consented patients (>18yo) on ventilatory support in the ICU at OHSU

Exclusion Criteria:

* Patients with "severe respiratory distress" as defined by arterial pO2 of <60 mmHg on maximal FiO2 & optimal ventilator settings
* Patient with severe hemodynamic instability as defined by (a) receiving IV infusion of 2 or more pressors or inotropic medications (Levophed, vasopressin, phenylephrine, or epinephrine) & (b) MAP of <60 mmHg or SB <80 mmHg

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Decisionally impaired adults will be included as part of the trauma population. The study aims to enroll patients who require ventilation support therefore qualifying some patients as decisionally impaired. Prisoners and pregnant women are excluded. Individuals under the age of 18 will not be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Exhaled breath-based diagnostic platform for detecting ventilator-associated pneumonia (VAP) early in critically ill, mechanically ventilated patients. | Admission to discharge (up to 30 days)
  This platform leverages advanced breath sampling technology and a host-response-based assay to detect specific elevated neutrophil proteases during bacterial infections like VAP. The noninvasive approach provides a safer and more efficient alternative to methods like bronchoalveolar lavage (BAL). This approach can differentiate between bacterial colonization and active infection by capturing and analyzing exhaled breath, allowing clinicians to initiate more timely and targeted therapies, thereby improving patient outcomes and reducing the misuse of antibiotics.

SECONDARY OUTCOMES:
Evaluate the effects of antibiotic treatment over time | Admission to discharge (up to 30 days)
  By tracking the levels of specific host-response markers in exhaled breath, the approach can monitor the progression or resolution of infection in real time. This data will provide critical insights into whether antibiotic therapy is effectively reducing the infection or if adjustments to the treatment regimen are needed. This will help reduce the overuse of antibiotics, support the fight against antimicrobial resistance, and improve patient outcomes in ICUs.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be shared with other researchers who are interested in any secondary analysis of the study.
Supporting Information: Study Protocol, SAP
Time Frame: The study data will be available at the end of study enrollment and will only be available until primary study analysis is complete.